CLINICAL TRIAL: NCT00145431
Title: Phase 3, Multi-Center, Double-Blind, Randomized, Crossover Study Of The Efficacy, Safety, And Tolerability Of Fixed Combination Torcetrapib (Cp-529,414)/Atorvastatin, Compared With Atorvastatin Therapy Alone, And Fenofibrate Alone, In Subjects With Fredrickson Type III Hyperlipoproteinemia (Familial Dysbetalipoproteinemia).
Brief Title: Study To Evaluate The Effect Of Torcetrapib/Atorvastatin In Subjects With A Genetic Cholesterol Disorder.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A5091024
Record Dates: First submitted 2005-08-31; First posted 2005-09-05 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Hyperlipoproteinemia Type III
MeSH Terms: conditions — Hyperlipoproteinemia Type III | interventions — torcetrapib; Atorvastatin; Fenofibrate

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin
Drug: fenofibrate

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To evaluate the efficacy and safety of the lipid drug torcetrapib/atorvastatin in subjects with a rare genetically known disorder of high cholesterol and triglyceride levels.

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Familial Dysbetalipoproteinemia (Fredrickson Type III hyperlipoproteinemia)

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in LDL-C and non-HDL-C levels.

SECONDARY OUTCOMES:
Changes in other lipid and biomarker variable levels.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (21):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Pacific Palisades, California
  - Pfizer Investigational Site, Studio City, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Tripler Army Medical Center, Hawaii
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Portage, Michigan
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Canada (4):
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec